CLINICAL TRIAL: NCT06543186
Title: Effectiveness of Metaverse-Based Immersive Technology Intervention for Oral Health Education: A Quasi-Experimental Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Amirul Faiz bin Luai, Postgraduate Student, Universiti Teknologi Mara
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC/07/2023 (PG/MR/228)
Record Dates: First submitted 2024-07-26; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: metaverse; immersive technology; virtual reality
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be assigned to one of the intervention groups based on designated locations within their schools: the main hall for the conventional oral health education group, classrooms for the WhatsApp group, and the computer lab for the Meta-OHE group. The interventions will be administered simultaneously to all groups by trained and calibrated researchers to minimize study contamination. This simultaneous approach ensures that each group receives the intervention under comparable conditions, thereby enhancing the reliability and validity of the study outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional oral health education (Experimental): For the conventional oral health education, the trained and calibrated dentist will provide health education to the selected participants in this group by chalk and talk method, PowerPoint presentations, models and charts so that it can make the sessions more interactive. The duration of the session will be around 60-90 minutes. Pre-assessment will be taken prior to the lecture. Post assessment will be taken after the lecture to assess the oral health knowledge, practise and attitude.
  Interventions: Other: Oral health education lecture
- Oral health education via mHealth using WhatsApp (Experimental): For the oral health education intervention via mHealth, WhatsApp medium will be used to disseminate oral health educational material. Before the commencement of the study, the participants will be asked for their phone number in the respondent sheet and permission will be sought from both participants and their teachers and parents/guardians. Then, a WhatsApp group will be created consisting of the selected participants for this intervention. The participants in WhatsApp group will further receive WhatsApp instant messages. These participants will grouped and placed in class. These messages will be sent in both Malay and English language. The duration of the session will be around 60-90 minutes. Pre-assessment will be taken prior to the dissemination of oral health education on WhatsApp. Post assessment will be taken afterwards to assess the oral health knowledge, practise and attitude.
  Interventions: Other: Oral health education via mHealth on WhatsaApp
- Metaverse platform called Metaverse for Oral Health Education (Meta-OHE) (Experimental): For oral health education intervention via Meta-OHE, it will be done via computer in a computer lab. The participants will be gathered in their school's computer lab with the health of the teacher. Participants will be assigned a computer to each of them. Then, they will be asked to sign in into Mitoworld platform using their respective email address on https://mitoworld.io/world/w/2808/meta-ohe to access Meta-OHE. They will be asked to enter the Meta-OHE portal. The students are permitted to freely explore and follow the instruction to visit each section of the Meta OHE and interact with each other. They will also be assigned a few tasks for them to complete on the platform to ensure all the oral health education materials are being covered. The duration of the session will be around 60-90 minutes. Pre-assessment will be taken prior to their access to Meta-OHE. Post assessment will be taken afterwards to assess the oral health knowledge, practise and attitude.
  Interventions: Other: Oral health education via Metaverse platform on Meta-OHE

INTERVENTIONS:
Other: Oral health education lecture — Conventional oral health education will be given by trained and calibrated dentists.
  Arms: Conventional oral health education
Other: Oral health education via mHealth on WhatsaApp — For the oral health education intervention via mHealth, WhatsApp medium will be used to disseminate oral health educational material
  Arms: Oral health education via mHealth using WhatsApp
Other: Oral health education via Metaverse platform on Meta-OHE — For oral health education intervention via Meta-OHE, it will be done via computer.
  Arms: Metaverse platform called Metaverse for Oral Health Education (Meta-OHE)

SUMMARY:
To evaluate the effectiveness of pre- and post-intervention of oral health education using three interventions (conventional methods, mHealth, and the Metaverse platform) on the oral health status, knowledge, practices, and attitudes among secondary school students in Malaysia.

DETAILED DESCRIPTION:
Background: In the last couple of years, the reach of the Internet is leading the world into a unique virtual dimension. Immersive technologies such as virtual reality (VR), augmented reality (AR), mixed reality (MR), extended reality (XR), and metaverse offer diverse virtual experiences and are gaining attention for their supportive role in addressing general health and oral health concerns. Dwivedi et al., in 2022, discussed and set out the potential research agenda in the metaverse in education and health. The metaverse environment offers users an immersive component and experience compared to the traditional environment . According to Locurcio, oral health education and promotion can be provided virtually to target groups and communities through public or private health sector metaverse software for public benefits. Due to no additional cost or limitation in the number of participants, it can educate multiple target groups by providing different sessions from anywhere in the world. These can benefit schoolchildren, teachers, and caregivers. Due to the immersive and interactive nature, the creation of safe and controlled environments and adaptation to the learners' characteristics, immersive technologies and metaverse specifically can facilitate and increase the inclusion of students in educational activities. Hence, the metaverse in oral health promotion and education can revolutionise how people learn, practise, and maintain good oral health. It can also make oral health information more accessible, engaging, and practical, ultimately leading to a positive behavioural change in oral health. Currently, virtual oral health education is often delivered through online platforms like social media, Zoom, Google Meet, and Microsoft Teams. In the future, individually customised oral health education will likely utilise more natural-feeling and immersive platforms, such as the metaverse. The development of metaverse platforms is intricate and context-specific and necessitates input from various relevant stakeholders. Few studies on creating health promotion applications have demonstrated that youth have distinct preferences for digital interventions compared to adults.

Aim: To evaluate the effectiveness of pre- and post-intervention of oral health education using three interventions (conventional methods, mHealth, and the Metaverse platform) on the oral health status, knowledge, practices, and attitudes among secondary school students in Malaysia.

Participants: Secondary school students from identified semi-government school in Malaysia.

Study risk: Participation to this study will not possess any potential risk, and the risk is minimal. Partcipants are free to decline to answer any of the questions that they feel uncomfortable with.

Benefits of the study: There may or may not be any benefits to the participants.

The study involves 15-16 years old adolescents enrolling in a semi-government school in Malaysia which will be divided into three groups that receive three interventions simultaneously at the same time and place (conventional methods, mHealth, and the Metaverse platform)

Duration of the study: Expected to be within six (months) from 1/05/2024 - 31/12/2024

Funding: This research received no external funding.

Conflicts of Interest: The authors declare no conflict of interest.

Ethical Policy and Review Board Statement: The study was approved by the UiTM Faculty of Dentistry Research Ethics Committee (FRC) [REC/07/2023 (PG/MR/228)]. Permission was granted from the Majlis Amanah Rakyat to use Maktab Rendah Sains MARA (MRSM) schools as study sites [MARA.600-6/1/6 JLD2 (56)].

ELIGIBILITY:
Inclusion Criteria:

1. aged 15-16 years old in 2024
2. voluntarily wish to participate in the research with consent from their legal guardians
3. enrolled in a co-education school (providing education to both boys and girls)
4. willing to commit to the program
5. can understand both Malay and English
6. participating schools must possess the necessary computer facilities to facilitate this aspect of the study

Exclusion Criteria:

1. aged less or more than 15-16 years old in 2024
2. not voluntarily wish to participate in the research with consent from their legal guardians
3. not enrolled in a co-education school (providing education to both boys and girls)
4. not willing to commit to the program
5. can't understand both Malay and English
6. participating schools does not possess the necessary computer facilities to facilitate this aspect of the study

Ages: 15 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Oral health knowledge | Pre-intervention (baseline) and immediately after the intervention
  Level of oral health knowledge. Descriptive, association and correlation
Oral health practise | Pre-intervention (baseline) and immediately after the intervention
  Level of oral health practise. Descriptive, association and correlation
Oral health attitude | Pre-intervention (baseline) and immediately after the intervention
  Level of oral health attitude. Descriptive, association and correlation

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Maktab Rendah Sains MARA Bentong, MRSM Bentong, Bentong, Pahang
  - Faculty of Dentistry, Universiti Teknologi MARA, Sungai Buloh, Selangor

IPD SHARING:
Plan to Share IPD: Yes
All the information obtained in this study ARE STRICTLY CONFIDENTIAL will be kept and handled in a confidential manner, in accordance with applicable laws and/or regulations. When publishing or presenting the study results, the participants' identity will not be revealed without your expressed consent. Individuals involved in this study, qualified monitors and auditors, and governmental or regulatory authorities may inspect the study data, where appropriate and necessary. All the data will be kept in a password protected folder that only can be access by the researcher. To obtain such information, a formal email need to be sent to the researcher at amirulfaiz2308@gmail.com (personal email) or 2022622294@student.uitm.edu.my (university email). Stored in non-publicly available repository, Available on request, Published as a supplement to the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years